CLINICAL TRIAL: NCT04328233
Title: Impact of Time-Restricted Eating on Metabolic and Neuroendocrine Homeostasis, Inflammation and Oxidative Stress in Patients With Metabolic Syndrome: the TREMNIOS Pilot Clinical Trial
Brief Title: Impact of Time-Restricted Eating on Metabolic Homeostasis, Inflammation and Oxidative Stress in Metabolic Syndrome
Acronym: TREMNIOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nicolaus Copernicus University (Other)
Collaborators: Salk Institute for Biological Studies (Other); University of California, San Diego (Other); Center for Obesity and Metabolic Disorders Treatment Bydgoszcz (Unknown)
Responsible Party: Principal Investigator, Iwona Swiatkiewicz, MD, PhD, FESC, Professor of Medicine, Nicolaus Copernicus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCU CM IRB 107/2019
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Syndrome; Overweight or Obesity; PreDiabetes; Weight Loss; Quality of Life
Keywords: Time-Restricted Eating; Circadian Rhythm; Glucose Homeostasis; Fasting; Metabolic Syndrome; Overweight; Obesity; PreDiabetes; Weight Loss; Metabolic Homeostasis; Neuroendocrine Biomarkers; Inflammation; Oxidative Stress
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Prediabetic State; Weight Loss; Intermittent Fasting; Fasting; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Time-Restricted Eating

INTERVENTIONS:
Behavioral: Time-Restricted Eating — Participants will reduce the amount of time they eat to 10 hours per day over a 12-week monitored intervention followed by a 12-week self-directed intervention and will log their dietary intake using a smartphone application (mCC app). The participants will select a 10-h eating window that best suits their lifestyle. All food/beverages except water must be consumed within the time-interval. No further dietary restrictions will be applied. The participants will be provided with behavioral nutritional counseling by a dietician.

SUMMARY:
The main purpose of the clinical trial is to determine the health impact of a dietary intervention known as time-restricted eating (TRE) in patients with metabolic syndrome (defined as the presence of elevated fasting plasma glucose and two or more of the following criteria: increased waist circumference, elevated fasting plasma triglycerides, reduced high-density lipoprotein-cholesterol, elevated blood pressure) and self-reported dietary intake of ≥14 hours per day. Participants will reduce the amount of time they eat to 10 hours per day over a 12-week monitored intervention followed by a 12-week self-directed intervention and will log their dietary intake using a smartphone application (myCircadianClock (mCC) app). Glucose homeostasis (blood glucose levels will be monitored continuously for 2 weeks at the baseline, at the end of the monitored intervention, and at the end of the self-directed intervention using a continuous glucose monitor), and other metabolic, neuroendocrine, inflammatory and oxidative stress/antioxidant defense biomarkers, body weight and composition, blood pressure, heart rate, sleep and activity (using mCC app), personal sense of wellness and dietary timing (using health questionnaires) will be evaluated at the baseline, at the end of the monitored intervention, and at the end of the self-directed intervention.

DETAILED DESCRIPTION:
Metabolic syndrome occurs in approximately 30% of adults and is associated with increased risk of cardiovascular disease and type 2 diabetes. Circadian rhythm disruption due to lifestyle including erratic eating patterns may lead to metabolic and neuroendocrine dysfunction, inflammation, oxidative stress, and cardiometabolic diseases. Maintaining a daily rhythm of eating and fasting cycles sustains a robust circadian rhythm which improves cellular bioenergetics and metabolism. Recent studies support the notion that restricting a period of food intake to 8-12 hours a day (time-restricted eating, TRE) can prevent and reverse obesity and metabolic dysfunction.

The main purpose of the clinical trial is to determine the health impact of TRE in patients with metabolic syndrome (defined as the presence of elevated fasting plasma glucose and two or more of the following criteria: increased waist circumference, elevated fasting plasma triglycerides, reduced high-density lipoprotein-cholesterol, elevated blood pressure) and self-reported dietary intake of ≥14 hours per day. Participants will reduce the amount of time they eat to 10 hours per day over a 12-week monitored intervention followed by a 12-week self-directed intervention and will log their dietary intake using a smartphone application (myCircadianClock (mCC) app, developed by the Salk Institute for Biological Studies). The participants will select a 10-h eating window that best suits their lifestyle. All food/beverages except water must be consumed within the time-interval. No further dietary restrictions will be applied. The participants will be provided with behavioral nutritional counseling by a dietician. Glucose homeostasis (blood glucose levels will be monitored continuously for 2 weeks at the baseline, at the end of the monitored intervention, and at the end of the self-directed intervention using a continuous glucose monitor), and other metabolic, neuroendocrine, inflammatory and oxidative stress/antioxidant defense biomarkers, body weight and composition, blood pressure, heart rate, sleep and activity (using mCC app), personal sense of wellness and dietary timing (using health questionnaires) will be evaluated at the baseline, at the end of the monitored intervention, and at the end of the self-directed intervention. The investigators will assess for compliance with TRE using mCC app.

ELIGIBILITY:
Inclusion Criteria:

1. Metabolic syndrome, defined as the presence of elevated fasting plasma glucose ≥ 100 mg/dL and two or more of the following criteria:

   Elevated waist circumference: ≥ 102 cm in men, ≥ 88 cm in women; Fasting plasma triglycerides ≥ 150 mg/dL (or on drug treatment for elevated triglycerides); Reduced High-density lipoprotein (HDL)-cholesterol < 40 mg/dL in men, < 50 mg/dL in women (or drug treatment for reduced HDL-cholesterol); Elevated blood pressure, Systolic blood pressure ≥ 130 mm Hg and/or diastolic blood pressure ≥ 85 mm Hg (or drug treatment for hypertension).
2. BMI > 25
3. Duration of eating period ≥ 14 hours/day.
4. Own a Smartphone with Apple Operating System (OS) or Android OS.

Exclusion Criteria:

1. Diagnosis of diabetes.
2. Pregnant or lactating women.
3. Active smoking or illicit drug use or history of treatment for alcohol abuse.
4. Shift work.
5. Caregivers for dependent requiring nocturnal care.
6. Planned travel over time zones during the study period.
7. History of major adverse cardiovascular event within the past 1 year (acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack) or current uncontrolled arrhythmia.
8. Uncontrolled medical conditions due to rheumatologic, hematologic, oncologic, infectious, gastrointestinal, psychiatric, nephrological, or endocrine diseases.
9. Known history of an eating disorder.
10. Currently enrolled in a weight-loss or weight-management program.
11. Special or prescribed diet for other reasons (e.g. Celiac disease).
12. Current treatment with antidepressants, medications affecting appetite, or immunosuppression.
13. History of bariatric surgery.
14. A score of > 16 on the Epworth Sleepiness Scale.
15. Depression determined by the Beck Depression Inventory.
16. Failure to use the smartphone app for documentation during a 2-week baseline period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline and after 14 weeks
  Body weight (kg) as measured in fasted state on a digital scale
Change in fasting glucose concentration | Baseline and after 14 weeks
  Fasting plasma glucose concentration (mg/dl)

SECONDARY OUTCOMES:
Body weight | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Body weight (kg) as measured in fasted state on a digital scale
Body mass index | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Body mass index (kg/m^2) as calculated from body weight (kg) and height (m)
Mean glucose | Changes from baseline. Measured at baseline, after 14 weeks, and after 26 weeks
  Glucose levels as measured by continuous glucose monitor (mg/dl) for 14 days at baseline, after 14 weeks, and after 26 weeks
Fasting glucose | Changes from baseline. Measured at baseline, after 14 weeks, and after 26 weeks
  Fasting glucose levels as measured by continuous glucose monitor (mg/dl) for 14 days at baseline, after 14 weeks, and after 26 weeks
Lipids | Changes from baseline. Measured in the blood in the fasted state at baseline, after 14 weeks, and after 26 weeks
  Fasting blood concentrations of lipids: total cholesterol (mg/dl), LDL cholesterol (mg/dl), HDL cholesterol (mg/dl), and triglycerides (mg/dl)
Fat mass | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Fat mass percentage (%) as measured by body composition analyzer (using bioelectric impendence technology)
HbA1c | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  HbA1c (%) assessed from blood samples
Metabolic and neuroendocrine biomarkers | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Fasting blood concentrations of metabolic and neuroendocrine biomarkers including but not limited to: free fatty acids, insulin, insulin-like growth factor-1, resistin, adiponectin, leptin, visfatin, irisin, ghrelin, omentin-1, and melatonin
Inflammatory biomarkers | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Fasting blood concentrations of inflammatory biomarkers including but not limited to: high sensitivity C-reactive protein, interleukin-6, interleukin-8, interleukin-10, tumor necrosis factor-α, tumor growth factor-β1, growth/differentiation factor 15
Oxidative stress/antioxidant defense biomarkers | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Fasting blood concentrations of oxidative stress/antioxidant defense biomarkers including but not limited to: superoxide dismutase-1, catalase, glutathione peroxidase, oxidized LDL, thiobarbituric acid reactive substances, conjugated dienes, malondialdehyde, 4-hydroxynonenal, vitamin A, and vitamin E
Waist circumference | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Waist circumference (cm) as measured using tape measure
Blood pressure | Changes from baseline. Fasted state at baseline, after 14 weeks, and after 26 weeks
  Systolic and diastolic blood pressure (mmHg) measured under resting and fasting conditions
Heart rate | Changes from baseline. Measured at baseline, after 14 weeks, and after 26 weeks
  Heart rate (bpm) measured under resting conditions during measurements of blood pressure
Energy intake | Registered at baseline, after 14 weeks, and after 26 weeks
  Energy intake (kcal/day) assessed from diet records
Timing of dietary intake | Changes from baseline. Registered at baseline, after 14 weeks, and after 26 weeks
  Timing of dietary intake (hh:mm) assessed from diet records and from the chrono-nutrition questionnaire
Self-reported sleepiness | Changes from baseline. Assessed at baseline, after 14 weeks, and after 26 weeks
  Self-reported sleepiness as assessed from the questionnaire the Epworth Sleepiness Scale
Self-reported sleep quality | Changes from baseline. Assessed at baseline, after 14 weeks, and after 26 weeks
  Self-reported sleep quality as assessed from the questionnaire Pittsburgh Sleep Quality Index
Self-reported chronotype | Changes from baseline. Assessed at baseline, after 14 weeks, and after 26 weeks
  Self-reported chronotype as assessed from the Munich Chronotype Questionnaire
Self-reported overall health and wellbeing | Changes from baseline. Assessed at baseline, after 14 weeks, and after 26 weeks
  Self-reported overall health and wellbeing as assessed from the questionnaire Self-reported health (SF-36 health survey)
Duration of eating period | Changes from baseline. Assessed at baseline, after 14 weeks, and after 26 weeks
  Duration from the first to last caloric intake over 24-hour cycle, collected via the smartphone app (mCC app)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Swiatkiewicz, MD, PhD, Principal Investigator — Nicolaus Copernicus University, Collegium Medicum Bydgoszcz
Locations (1):
- Nicolaus Copernicus University, Collegium Medicum Bydgoszcz, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaix A, Zarrinpar A, Miu P, Panda S. Time-restricted feeding is a preventative and therapeutic intervention against diverse nutritional challenges. Cell Metab. 2014 Dec 2;20(6):991-1005. doi: 10.1016/j.cmet.2014.11.001. PMID 25470547
- [Background] Gill S, Le HD, Melkani GC, Panda S. Time-restricted feeding attenuates age-related cardiac decline in Drosophila. Science. 2015 Mar 13;347(6227):1265-9. doi: 10.1126/science.1256682. PMID 25766238
- [Background] Panda S. Circadian physiology of metabolism. Science. 2016 Nov 25;354(6315):1008-1015. doi: 10.1126/science.aah4967. PMID 27885007
- [Background] Pot GK, Almoosawi S, Stephen AM. Meal irregularity and cardiometabolic consequences: results from observational and intervention studies. Proc Nutr Soc. 2016 Nov;75(4):475-486. doi: 10.1017/S0029665116000239. Epub 2016 Jun 22. PMID 27327128
- [Background] Gill S, Panda S. A Smartphone App Reveals Erratic Diurnal Eating Patterns in Humans that Can Be Modulated for Health Benefits. Cell Metab. 2015 Nov 3;22(5):789-98. doi: 10.1016/j.cmet.2015.09.005. Epub 2015 Sep 24. PMID 26411343
- [Background] Sulli G, Manoogian ENC, Taub PR, Panda S. Training the Circadian Clock, Clocking the Drugs, and Drugging the Clock to Prevent, Manage, and Treat Chronic Diseases. Trends Pharmacol Sci. 2018 Sep;39(9):812-827. doi: 10.1016/j.tips.2018.07.003. Epub 2018 Jul 27. PMID 30060890